CLINICAL TRIAL: NCT03568617
Title: Repetitive Transcranial Magnetic Stimulation for the Prevention Treatment of Chronic Migraine: a Single Arm Study
Brief Title: rTMS for the Prevention Treatment of CM: a Single Arm Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rTMSCM-PUMCH
Record Dates: First submitted 2018-06-04; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Chronic Migraine
Keywords: Transcranial Magnetic Stimulation; Migraine Disorders; Prophylaxis; Treatment Outcome; Brain
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS group (Experimental)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — The subjects will receive 20 trains of 100 stimuli each delivered at 10 Hz and 80% of MT over the left MC (M1), 3 days a week, for 4 weeks.

SUMMARY:
We design this pilot, single arm study to explore the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) for the treatment of chronic migraine. The hypothetical control group is pooled sham group in latest meta-analysis. We expect a significant improvement of the outcome measures during and after the treatment as compared to the hypothetical control group.

DETAILED DESCRIPTION:
After a 28-day prospective baseline period using a headache diary to record headache symptoms and any abortive medications used, subjects who meet diagnostic criteria for chronic migraine and don't meet the exclusion criteria will receive rTMS for 4 weeks. The outcome measure will be evaluated at 4 weeks. During the whole trial period, any adverse events are requested to be recorded in the headache diary for analyses. The primary outcome is 50% reduction in the number of days with headache. 50% reduction as assessed by migraine days, moderate/severe headache days, the mean VRS, and conversion to episodic migraine, SGIC, the change from baseline HALT-28, HIT-6, and MSQ v2.1, are used as secondary outcome measures for exploring other benefits associated with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the diagnostic criteria for chronic migraine according to the International Classification of Headache Disorders, 3rd edition.
* The duration of chronic migraine ≥ 6 months.
* age range of 18 - 65 years old

Exclusion Criteria:

* Secondary headaches except MOH
* any change of the prophylaxis or the analgesic drug strategy during the baseline and follow-up period
* structural brain lesions
* seizures
* severe systemic disease
* TMS contraindications (such as metal implants)
* psychosis
* severe depression or anxiety
* drug or alcohol dependence
* pregnancy
* participating in other experiments at the same time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
50% reduction in the Number of Days with Headache | at 4 weeks
  A Headache day is defined as a day with a headache that lasts at least 4 hours.

SECONDARY OUTCOMES:
50% reduction in the Number of Migraine Days | at 4 weeks
  A migraine day is defined as a day with a headache that lasts at least 4 hours; meets ICHD-III criteria C and D for migraine without aura (1.1), B and C for migraine with aura (1.2), or ICHD-III criteria for probable migraine (1.6); or a day with a headache that is successfully treated with a triptan, ergotamine, or other migraine-specific acute medication.
50% reduction in the Number of Moderate/Severe Headache Days | at 4 weeks
  A moderate/severe headache day is defined as a day with moderate or severe pain that lasts at least 4 hours or a day with a headache that is successfully treated by an acute headache medication.
Conversion to episodic migraine | at 4 weeks
  Defined as the proportion of subjects with fewer than 14 migraine or headache days per 4 weeks.
The Subject's Global Impression of Change (SGIC) | at 4 weeks
  Global impression of change was scored using a 7-point scale for each instrument, ranging from 1 (very much improved) to 7 (very much worse), with a 4-week recall period. We'll estimate the proportion of patients who reported any improved (very much improved, much improved, minimally improved).
Change from Baseline HALT-28 (Headache-Attributed Lost Time - 28 days) | at baseline and 4 weeks
  HALT-30 is closely based on the first five questions of MIDAS, developed by RB Lipton and WF Stewart. We modify the time interval to capture migraine-related disability with a 4-week recall period.
Change from Baseline HIT-6 (Headache Impact Test-6) | at baseline and 4 weeks
  HIT-6 is for capturing migraine-related disability with a 4-week recall period.
Change from Baseline MSQ v2.1 (the Migraine-Specific Quality of Life questionnaire v2.1) | at baseline and 4 weeks
  To evaluate the change in quality of life related to chronic migraine with a 4-week recall period.
50% reduction as assessed by the mean VRS | at 4 weeks
  Subjects will be instructed to record the pain intensity of each day using 11-point Visual Rating Scale (VRS). The mean VRS is defined as the mean of the maximum VRS of each day with a 4-week period.

REFERENCES:
- [Background] Lan L, Zhang X, Li X, Rong X, Peng Y. The efficacy of transcranial magnetic stimulation on migraine: a meta-analysis of randomized controlled trails. J Headache Pain. 2017 Aug 22;18(1):86. doi: 10.1186/s10194-017-0792-4. PMID 28831756
- [Background] Shehata HS, Esmail EH, Abdelalim A, El-Jaafary S, Elmazny A, Sabbah A, Shalaby NM. Repetitive transcranial magnetic stimulation versus botulinum toxin injection in chronic migraine prophylaxis: a pilot randomized trial. J Pain Res. 2016 Oct 7;9:771-777. doi: 10.2147/JPR.S116671. eCollection 2016. PMID 27785091
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] Steiner TJ, Lipton RB; Lifting The Burden: The Global Campaign against Headache. The Headache-Attributed Lost Time (HALT) Indices: measures of burden for clinical management and population-based research. J Headache Pain. 2018 Feb 2;19(1):12. doi: 10.1186/s10194-018-0837-3. PMID 29396646